CLINICAL TRIAL: NCT06278467
Title: Frequency of Cognitive Dysfunction and Related Factors in Patients With Chronic Low Back Pain
Brief Title: Frequency of Cognitive Dysfunction in Patients With Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ramazan Yılmaz, Assist Prof (MD), Konya Beyhekim Training and Research Hospital
Other Study IDs: KonyaBeyhekimTRH2023
Record Dates: First submitted 2024-02-05; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cognitive Dysfunction; Low Back Pain
Keywords: cognitive dysfunction; low back pain; Chronic pain
MeSH Terms: conditions — Cognitive Dysfunction; Low Back Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with chronic low back pain: Consecutive patients over the age of 60, diagnosed with CBP, who have been suffering from low back pain for at least 6 months (n=57 )
  Interventions: Diagnostic Test: visual pain scale (VASpain/fatigue), Beck depression index (BDI),; Diagnostic Test: Pain catastrophizing scale, sleep quality with a single Likert type question in the Pittsburgh questionnaire; Diagnostic Test: Roland Morris Disability Questionnaire, quality of life with Short Form-36 ( SF-36),; Diagnostic Test: Montreal Cognitive Assessment Scale (MOCA); Standard Mini mental test (SMMT)
- Healtyh control: Healthy control with compatible sociodemographic characteristics (n=50)
  Interventions: Diagnostic Test: visual pain scale (VASpain/fatigue), Beck depression index (BDI),; Diagnostic Test: Pain catastrophizing scale, sleep quality with a single Likert type question in the Pittsburgh questionnaire; Diagnostic Test: Roland Morris Disability Questionnaire, quality of life with Short Form-36 ( SF-36),; Diagnostic Test: Montreal Cognitive Assessment Scale (MOCA); Standard Mini mental test (SMMT)

INTERVENTIONS:
Diagnostic Test: visual pain scale (VASpain/fatigue), Beck depression index (BDI), — VAS (0-10)
Diagnostic Test: Pain catastrophizing scale, sleep quality with a single Likert type question in the Pittsburgh questionnaire — PCS (Pain catastrophizing scale); sleep quality with a single Likert type question in the Pittsburgh questionnaire (0-3)
Diagnostic Test: Roland Morris Disability Questionnaire, quality of life with Short Form-36 ( SF-36), — functional disability level with Roland Morris Disability Questionnaire, quality of life with Short Form-36 ( SF-36)
Diagnostic Test: Montreal Cognitive Assessment Scale (MOCA); Standard Mini mental test (SMMT) — cognitive status was measured by Montreal Cognitive Assessment Scale (MOCA) and Standard Mini mental test (SMMT)

SUMMARY:
This study evaluates cognitive dysfunction status and related factors in patients with chronic low back pain over the age of 60.

DETAILED DESCRIPTION:
The study was designed as prospective, cross-sectional and hospital-based. 55 consecutive patients over the age of 60, diagnosed with CBP, who have been suffering from low back pain for at least 6 months, and a similar number of healthy volunteers (control) in terms of age and gender, who applied to the Physical Medicine and Rehabilitation outpatient clinic of Konya Beyhekim Training and Research Hospital, will be included in the study. Patients will be included in this cross-sectional, survey-type research after their compliance with the inclusion criteria is meticulously determined as a result of anamnesis and physical examination.

Detailed histories of all participants will be taken and detailed physical examinations will be performed. Sociodemographic and clinical characteristics of the participants, such as age, gender, height, weight, educational status, marriage status, duration of illness, and employment status, will be recorded.

Patients will be asked some survey-type questions in a decent environment. Patients' pain and fatigue levels were measured by the visual pain scale (VAS), their emotional states by the Beck depression scale (BDI) and Pain catastrophizing scale, their functional disability level by the Roland Morris Disability Questionnaire, and their sleep quality by the single Likert type question in the Pittsburgh questionnaire. Quality of life will be evaluated with Short Form-36 (SF-36), and their cognitive status will be evaluated with Standard Mini mental test (SMMT) and Montreal cognitive assessment scale (MOCA).MOCA, mini mental test and mood tests are administered by a professional psychologist experienced in the application of these scales.

ELIGIBILITY:
Inclusion Criteria:

Being over 60 years old Having a history of low back pain lasting more than 6 months and being diagnosed with CBP Having pain of at least 3 intensity according to VAS

Exclusion Criteria:

Those under 60 years of age

* Those with neurological deficits
* Those with inflammatory low back pain
* Those with rheumatic diseases such as fibromyalgia, polymyalgia rheumatica, ankylosing spondylitis, rheumatoid arthritis
* Having undergone surgery in the lumbar region within the last 6 months
* Those with widespread pain, those with significant pain in another anatomical location (e.g. gonarthrosis)
* Those who use drugs or substances (alcohol, drugs, etc.) that may cause cognitive impairment
* Those with known neurological diseases such as cerebrovascular disease, MS, Parkinson's, dementia
* Those with major psychiatric illness
* Those with communication problems
* Those who have started psychiatric medical treatment within the last three months
* Those with significant hearing or vision problems
* Those with a history of uncontrolled systemic disease (cardiovascular, pulmonary, hepatic, renal, hematological, endocrine, etc.)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those with chronic low back pain over the age of 60 and healthy controls. Patients were included in the study according to the inclusion and exclusion criteria and on a voluntary basis.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Scale (MOCA) | 2022-2024
  minimum and maximum values: 0 - 30, and higher scores mean a better outcome.
Standard Mini mental test (SMMT) | 2022-2024
  minimum and maximum values: 0 -30, and higher scores mean a better outcome.
Short Form-36 ( SF-36) | 2022-2024
  minimum and maximum values: 0 -100, and higher scores mean a better outcome.
Beck depression scale (BDI) | 2022-2024
  minimum and maximum values: 0 -63, and higher scores mean a worse outcome.
Roland Morris Disability Questionnaire | 2022-2024
  minimum and maximum values: 0 - 24, and higher scores mean a worse outcome
A single Likert type question in the Pittsburgh questionnaire (Sleep quality) | 2022-2024
  minimum and maximum values: 0 - 3, and higher scores mean a better outcome
VAS pain and VAS fatigue | 2022-2024
  VAS minimum and maximum values: 0 - 10, and higher scores mean a worse outcome
Pain catastrophizing scale | 2022-2024
  minimum and maximum values: 0 - 52, and higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Konya Beyhekim Training and Research Hospital, Konya, Selçuklu
  - University of Health Sciences, Konya Beyhekim Training and Research Hospital, Department of Physical Medicine and Rehabilitation, Konya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berryman C, Stanton TR, Jane Bowering K, Tabor A, McFarlane A, Lorimer Moseley G. Evidence for working memory deficits in chronic pain: a systematic review and meta-analysis. Pain. 2013 Aug;154(8):1181-96. doi: 10.1016/j.pain.2013.03.002. Epub 2013 Mar 14. PMID 23707355
- [Background] Corti EJ, Gasson N, Loftus AM. Cognitive profile and mild cognitive impairment in people with chronic lower back pain. Brain Cogn. 2021 Jul;151:105737. doi: 10.1016/j.bandc.2021.105737. Epub 2021 May 1. PMID 33945940